CLINICAL TRIAL: NCT04107051
Title: Nalmefene Hydrochloride Hydrate Tablets 10mg Specified Drug-use Results Survey (the Safety and the Prognosis After Achieving Reduced Alcohol Intake)
Brief Title: Post-Marketing Surveillance Study of Nalmefene Hydrochloride Hydrate in Patients with Alcohol Dependence
Status: Completed | Type: Observational
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: 339-101-00015
Record Dates: First submitted 2019-09-24; First posted 2019-09-27 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-02

CONDITIONS: Alcohol Dependence
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Nalmefene Hydrochloride Hydrate — Oral administration of nalmefene hydrochloride hydrate

SUMMARY:
The purpose of this study is to investigate the safety and the prognosis after achieving reduced alcohol intake in patients with alcohol dependence who received treatment for the reduction of alcohol intake in the routine clinical setting in Japan.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Alcohol Dependence
* Must agree to follow-up during the first year of prescription and publication of survey results
* Patients whose goal of treatment for Alcohol Dependence is to reduce alcohol consumption
* Patients receiving psychosocial treatment aiming to promote treatment adherence and reduction of alcohol consumption
* Patients who have chronic heavy drinking
* Patients who have confirmed that they are willing to receive treatment to reduce their alcohol consumption

Exclusion Criteria:

* Patients who has ever been treated with nalmefene hydrochloride hydrate
* Patients who are contraindicated

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with alcohol dependence who are planned to be newly started on nalmefene hydrochloride hydrate for the treatment of reduction of alcohol consumption.
Sampling Method: Non-Probability Sample
Enrollment: 533 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2023-02-07 (Actual); Study Completion 2024-02-06 (Actual)

PRIMARY OUTCOMES:
Alcohol Use Disorders Identification Test-Consumption(AUDIT-C) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Yasuhiko Fukuta, PhD, Study Director — Otsuka Pharmaceutical Co., Ltd.
Locations (1):
- Otsuka Pharmaceutical Co., Ltd., Osaka, Japan

IPD SHARING:
Plan to Share IPD: No